CLINICAL TRIAL: NCT06777706
Title: An Open-label Study to Assess the Safety and Efficacy of QD (Indigo Naturalis) Food Supplement for Induction of Remission in Pediatric Patients with Ulcerative Colitis
Brief Title: Open Label Study to Assess Safety & Efficacy of QD for Induction of Remission in Pediatric Patients with UC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QD
Record Dates: First submitted 2022-05-04; First posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Ulcerative Colitis; Inflammatory Bowel Diseases
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases | interventions — Qingdai compound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients receiving QD (Experimental): Patients will be receiving QD as oral capsules.
  Dosing of QD will be stratified based on body weight at time of enrollment:
  * 15-30kg: 500 mg/day (250 mg morning; 250 mg evening).
  * 30-40kg: 750 mg/day (500 mg morning; 250 mg evening).
  * >40kg: 1000mg/day (500 mg morning; 500 mg evening).
  If the patient fails to respond by week 3 to current dosing regimens (failure defined as <20 decrease in PUCAI and PUCAI>10), and if no safety concerns arise at week 3, dose will be increased, as following:
  * 15-30kg: 1000 mg/day (500 mg morning; 500 mg evening)
  * 30-40kg: 1500 mg/day (1000 mg morning; 500 mg evening)
  * >40kg: 2000mg/day (1000 mg morning; 1000 mg evening)
  Interventions: Dietary Supplement: QD (Qing Dai)

INTERVENTIONS:
Dietary Supplement: QD (Qing Dai) — Children age 4 years to 17.9 years with mild to moderate UC will receive QD and dosing will be stratified based on body weight at time of enrollment.

SUMMARY:
To date, there are no reports on the use of QD in pediatric patients with UC. There is a great need to increase the repertoire of anti-inflammatory interventions for remission induction, especially in children given the notorious side effects of steroids on growth. Importantly, no prescription is needed to acquire QD, as this is a food supplement that can be purchased over the counter. We wish to assess the efficacy and safety of QD as induction therapy in pediatric patients with mild-moderate active UC.

DETAILED DESCRIPTION:
This is a prospective open-label pilot study in two Pediatric IBD centers at Schneider Children's Medical Center of Israel and Share Zedek Medical Center. Pediatric UC patients at both participating centers will be screened during clinic visits for eligibility to participate in the study. Eligible patients are 4-17.9 years old, with at least one month history of UC, with mild to moderate active UC, defined by a PUCAI score of 10-60, despite current treatment. Normal liver enzymes obtained within one most prior to initiation of the study is required. The study will be presented to the families and once it is established that the patient fulfills the inclusion criteria, informed written consent will be obtained from the patient and parents.

Enrollment:

At enrolment patients will be examined and explicit clinical, medical and demographic data will be documented. PUCAI16 and TUMMY-UC (patient reported outcome developed specifically for pediatric UC patients17) scores will be determined. Extent of disease will be documented according to the last available colonoscopy, using the Montreal classification definitions (additional endoscopic evaluation is not required for the study). Laboratory work including CBC, albumin, AST, ALT, ESR and CRP. A stool sample will be obtained and kept at -800C for future analyses (see below). In addition, a baseline echocardiography will be performed to assess for PAH prior to initiation of QD (see below). Patients of child bearing potential will be advised to safeguard against pregnancy.

Following completion of enrollment and initial testing patients will receive QD (see dosing regimens below). QD will be provided as oral capsules. Patients who are not able to swallow the capsules will be instructed to open then and give it with yogurt/soft food. Patients will be instructed to continue taking their maintenance medication as prescribed by their treating physician throughout the entire study period, without any changes.

Day 3-4:

Patients will be contacted via telephone and questioned regarding any adverse effects, and specifically headaches, along with colitis-associated clinical features.

Week 3:

Patients will be seen in clinic, and will also be examined, as part of routine clinical care. Clinical data will be obtained, including PUCAI and TUMMY-UC. Prior to this visit, patients will complete blood work including CBC, chemistry panel and CRP. A stool sample will be collected at this clinic visit.

Week 6:

Patients will be seen in clinic, and will also be examined, as part of routine clinical care. Clinical data will be obtained, including PUCAI and TUMMY-UC. Patients will also complete prior to this visit blood work including CBC, chemistry panel and CRP. An additional stool sample will be obtained and kept at -80 degrees celsius for future analyses. Finally, a repeated echocardiography will be completed. At this timepoint, the study will be completed.

Termination visit:

If the study will be terminated prior to completion of the 6 weeks of QD therapy (see criteria below) the patient will be seen in clinic for a "termination visit". In this visit clinical data will be obtained, including PUCAI and TUMMY-UC. Patients will also complete prior to this visit blood work including CBC, chemistry panel and CRP. An additional stool sample will be obtained and kept at -80 degrees celsius. for future analyses.

At each study visit, patients of child bearing potential will be asked if they are pregnant.

ELIGIBILITY:
Inclusion Criteria:

1. Established diagnosis of UC for at least one month based on accepted criteria15.
2. Age 4-17.9 years old (inclusive).
3. Weight ≥ 15kg
4. PUCAI 10-60 at enrollment (reflecting mild-moderate UC).
5. If a patient is receiving oral 5-ASA, the dose must be stable for at least 4 weeks prior to inclusion.
6. If patient is receiving immunomodulator medication (azathioprine or 6- mercaptopurine), dose must be stable for at least 3 months prior to inclusion.
7. If a patient is on topical 5-ASA (suppositories or enema) the dose must be stable for at least 2 weeks prior to inclusion and will not be altered throughout the 6-week study period.
8. Negative stool culture, parasites and clostridium difficile testing.

Exclusion Criteria:

1. Acute severe colitis (PUCAI>65).
2. Patient with chronic renal or liver disease, hypertension, cardiovascular disease, cerebrovascular disease, chronic pancreatitis, diabetes mellitus, gallstone disease, previous malignancy, uncontrolled migraines or neurological disorders.
3. Abnormal liver enzymes (ALT, AST, GGT) X2 times upper normal limit.
4. Patients whose disease is confined to the rectum (i.e. proctitis).
5. Systemic steroid treatment at the time of enrollment (regardless of dose)
6. Prior or current treatment with biologic therapy or JAK inhibitor.
7. Patient with active infection.
8. Known immunodeficiency.
9. Known allergy to QD.
10. Pregnancy per questionnaire.

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Clinical remission at 6 weeks | Six weeks after the first dose of QD
  Rate of corticosteroid-free clinical remission at 6 weeks (defined as PUCAI<10) and a decrease in PUCAI score of at least 10.

SECONDARY OUTCOMES:
Rate of clinical response | Six weeks after the first dose of QD
  Rate of clinical response (PUCAI score decrease by 20 points or a decrease to less than 10) at week 6.
Calprotectin <250 mcg/g | Six weeks after the first dose of QD
  Rate of calprotectin <250 mcg/g at week 6.
Calprotectin decrease - week 6 | Six weeks after the first dose of QD
  Rate of calprotectin decrease at week 6 by >50% compared to baseline level
Rate of clinical remission | Three weeks after the first dose of QD
  Rate of clinical remission (PUCAI<10) at week 3.
Rate of clinical response | Three weeks after the first dose of QD
  Rate of clinical response (PUCAI score decrease by 20 points or a decrease to less than 10) at week 3.
Calprotectin <100 mcg/g - week 6 | Six weeks after the first dose of QD
  Rate of calprotectin <100 mcg/g at week 6.
PUCAI<10 and calprotectin <100 mcg/g | Six weeks after the first dose of QD
  Rate of PUCAI<10 and calprotectin <100 mcg/g at week 6.
Calprotectin decrease - week 3 | Three weeks after the first dose of QD
  Rate of calprotectin decrease at week 3 by >50% compared to baseline level.
Calprotectin <100 mcg/g - week 3 | Three weeks after the first dose of QD
  Rate of calprotectin <100 mcg/g at week 3.
PUCAI<10 and calprotectin <100 mcg/g - week 3 | Three weeks after the first dose of QD
  Rate of PUCAI<10 and calprotectin <100 mcg/g at week 3.
Rate of QD-associated adverse events | Six weeks after the first dose of QD
  Rate of QD-associated adverse events including but not limited to: PAH, elevation in liver enzymes, headaches.

CONTACTS AND LOCATIONS:
Overall Officials: Dotan Yogev, MD, Principal Investigator — Shaare Zedek Medical Center
Locations (2):
- Israel (2):
  - Shaare Zedek Medical Center - The Juliet Keidan Institute of Paediatric Gastroenterology and Nutrition, Jerusalem
  - Schneider Children's Medical Center, Petah Tikva